CLINICAL TRIAL: NCT00820651
Title: Efficacy and Safety of Diamel, a Nutritional Supplement, in Patients With Nonalcoholic Steatohepatitis. A Randomized and Double Blind Controlled Study
Brief Title: Efficacy and Safety of Diamel in Patients With Nonalcoholic Steatohepatitis
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Catalysis SL (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: DIAMEL_NASH-09
Record Dates: First submitted 2009-01-09; First posted 2009-01-12 (Estimated); Last update posted 2012-04-26 (Estimated); Status verified 2012-04

CONDITIONS: Nonalcoholic Steatohepatitis; Insulin Resistance
Keywords: Nonalcoholic steatohepatitis; Insulinresistance; Diet and exercise; Nutritional supplement; Nonalcoholic fatty liver disease; Lifestyle modifications
MeSH Terms: conditions — Non-alcoholic Fatty Liver Disease; Insulin Resistance; Motor Activity | interventions — Dietary Supplements

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Placebo (Placebo Comparator)
  Interventions: Other: Placebo and lifestyle counseling
- Diamel (Experimental)
  Interventions: Dietary Supplement: Diamel

INTERVENTIONS:
Dietary Supplement: Diamel — Diamel, a nutritional supplement, 2 oral pills (660 mg), every 8 hours, daily, during 52 weeks
  Other Names: Dietary supplement
  Arms: Diamel
Other: Placebo and lifestyle counseling — Hypocaloric diet of 1620 kcal daily (The dietary pattern will be distributed in carbohydrates 64%, fat 22% with <10% of saturated fatty acids and protein 14%, and exercise)
  Other Names: Placebo; Lifestyle modification
  Arms: Placebo

SUMMARY:
The purpose of the study is to evaluate whether the addition of Diamel, a nutritional supplement, to hypocaloric diet and exercise could improve the histological results (steatosis, necro-inflammatory activity and fibrosis), insulin resistance, aminotransferase levels and anthropometric measures in comparison with a placebo-controlled group with hypocaloric diet and exercise during 52 weeks of treatment in patients with nonalcoholic steatohepatitis.

ELIGIBILITY:
Inclusion Criteria:

* Histological diagnosis of steatohepatitis (minimal histological criteria for steatohepatitis include steatosis involving at least 5% of hepatocytes, lobular inflammation, and/or fibrosis)
* Age between 18 and 70 years
* Ability to provide informed consent
* Absence of significant alcohol ingestion (weekly ethanol consumption of less than 40 g)

Exclusion Criteria:

* Presence of other form of liver diseases (viral or autoimmune hepatitis, drug-induced liver disease, metabolic and hereditary liver disease and α-1 antitrypsin deficiency)
* Pregnancy or lactation
* Decompensated cirrhosis
* Presence of secondary cause of NAFL such as medications that induce steatosis (corticosteroids, estrogens, methotrexate, amiodarone, tamoxifen and calcium channel blockers) and gastrointestinal bypass surgery
* Pharmacological treatment with some potential benefit on NAFL including ursodeoxycholic acid, vitamin E, betaine, pioglitazone, rosiglitazone, metformin, pentoxifylline or gemfibrozil
* Fasting glucose levels greater than 250 mg per deciliter (13.3 mmolm per liter)
* Contraindication to liver biopsy
* Refusal to participate in the study
* Concomitant disease with reduced life expectancy
* Severe psychiatric conditions
* Drug dependence

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 158 (Actual)
Dates: Start 2009-11; Primary Completion 2012-04 (Actual); Study Completion 2012-04 (Actual)

PRIMARY OUTCOMES:
The histological improvement (steatosis, necro-inflammatory activity and fibrosis) at 52 weeks (end of the treatment) as compared with pre-treatment liver biopsy. | 52 weeks

SECONDARY OUTCOMES:
Insulinresistance levels (HOMA-IR) at 52 weeks (end of the treatment), Aminotransferase levels at 52 weeks (end of the treatment), Body weight, Body Mass Index and waist circumference at 52 weeks (end of the treatment) | 52 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Eduardo Vilar Gomez, Ph.D, Principal Investigator — National Institute of Gastroenterology
Locations (1):
- National Institute of Gastroenterology, Vedado, La Habana, Cuba

REFERENCES:
- [Result] Hernandez Yero JA, Vargas Gonzalez D. Utilidad de Diamel en pacientes con diabetes mellitus tipo 2 en tratamiento combinado con glibenclamida. Avances en Diabetología 23(1):284-290, 2007